CLINICAL TRIAL: NCT07275671
Title: A Case-Control Study of Gut and Vaginal Microbiota Differences Between Premature Ovarian Insufficiency Patients and Healthy Controls
Brief Title: Microbiome and Premature Ovarian Insufficiency
Status: Recruiting | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20250416ZJS004
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Premature Ovarian Insufficiency; Reproductive Health
Keywords: Premature Ovarian Insufficiency; Gut microbiome; Vaginal microbiome
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood, Stool, Urine, Vaginal swab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POI: Premature ovarian insufficiency
- CTL: Healthy control

SUMMARY:
This study investigates the differences in gut and vaginal microbiota between women with premature ovarian insufficiency (POI) and healthy volunteers. POI refers to the reduction in ovarian function before the age of 40, leading to irregular or absent menstruation and decreased estrogen levels, which can significantly affect women's reproductive and overall health. Recent research has suggested that gut microorganisms may influence the balance of steroid hormones through various metabolic pathways. Additionally, certain vaginal bacteria appear enriched in patients with POI, but whether these microorganisms directly impact ovarian function, and how, remains unclear. This study also seeks to address the underexplored role of fungi within the human microbiome. To comprehensively compare differences in gut and vaginal microbiota, the study will recruit 20 women with POI and 20 healthy controls. Both demographic and clinical information will be collected, along with biological samples including blood, urine, stool, and vaginal swabs.

DETAILED DESCRIPTION:
This project utilizes a case-control study design to systematically compare the microbiome profiles of women diagnosed with premature ovarian insufficiency (POI) and healthy controls. A total of 20 participants with POI and 20 age-matched healthy volunteers will be recruited. Biological samples collected will include blood, midstream urine, stool, and vaginal swab per participant. Blood samples will be obtained by licensed nurses; for menstruating women, samples are drawn during days 2-5 of the most recent cycle, while for those with amenorrhea or menopause, samples are taken at any time for serum hormone testing. Vaginal swab samples are collected by experienced gynecologists, avoiding collection during menstruation. Urine samples are self-collected by volunteers and immediately handed over to research staff for freezing, while stool samples are self-collected and sent to the laboratory staff by low-temperature shipping for prompt processing and storage. Both samples are collected outside of the menstrual period. Comprehensive baseline data will be obtained through questionnaires and electronic medical records by trained interviewers. This includes demographic details, lifestyle factors, reproductive and menstrual history, use of antibiotics and supplements, Kupperman Index (KMI), Hospital Anxiety and Depression Scale (HAD), and sleep quality assessments. All biosamples will be handled according to strict aseptic procedures, aliquoted and stored at -80°C for subsequent omics analyses. Data collection and quality control procedures will be overseen and maintained by the research team for long-term storage and analysis.

ELIGIBILITY:
Inclusion Criteria:

(For POI patients)

1. Women aged 20 to 40 years at screening visit.
2. Clinical diagnosis of premature ovarian insufficiency (based on diagnostic criteria: 25 < FSH ≤ 40 IU/L, reduced follicle count and abnormal follicle development by ultrasound).
3. Able to provide informed consent.

(For healthy volunteers)

1. Age (±2 years) and sex-matched healthy control individuals for each POI patient.
2. Able to provide informed consent.

Exclusion Criteria:

(For POI patients)

1. Family history of premature ovarian insufficiency.
2. Use of hormone therapy (such as HRT) within the past 6 months.
3. Serious illness (e.g., heart failure or malignancy).
4. Smoking more than 15 cigarettes per day or history of alcohol or drug addiction.
5. Inflammatory gastrointestinal diseases.
6. Chronic diseases that may affect the gut microbiota (e.g., diabetes, cirrhosis, or cardiovascular disease).
7. Blood or autoimmune diseases, or use of immunosuppressants in the past 3 months.
8. Use of antibiotics in the past 3 months before sample collection.
9. Chronic constipation.

(For healthy volunteers)

1. Have a history of infertility or recurrent miscarriage.
2. Pregnant or breastfeeding.
3. Use of hormone therapy (e.g., loratadine, oral contraceptives, etc.) within the past 6 months.
4. Inflammatory gastrointestinal diseases.
5. Smoking more than 15 cigarettes per day or history of alcohol or drug addiction.
6. Chronic diseases that may affect the gut microbiota (e.g., diabetes, cirrhosis, or cardiovascular disease).
7. Blood or autoimmune diseases, or use of immunosuppressants in the past 3 months.
8. Use of antibiotics in the past 3 months before sample collection.
9. Chronic constipation.
10. Participating in other clinical trials.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Study Population: All the participants should be residents living in East China.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome profiling | At enrollment
  The microbiome profile is analyzed based on stool samples in cases and controls.
Vaginal microbiome profiling | At enrollment
  The microbiome profile is analyzed based on vaginal swab samples.

SECONDARY OUTCOMES:
Blood and urine metabolomics profiling | At enrollment
  Proteomics profiles are analyzed based on blood samples and urine samples.
Fecal and serum metabolomics profiling | At enrollment
  Metabolomics profiles are analyzed based on blood samples and stool samples in cases and controls.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Changzheng Hospital, Shanghai
  - The Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided